CLINICAL TRIAL: NCT03569878
Title: A Comparative Effectiveness Trial of an Information Technology Enhanced Peer-Integrated Collaborative Care Intervention for US Trauma Care Systems
Brief Title: IT Enhanced Peer Integrated Collaborative Care for US Trauma Care Systems
Acronym: TSOS 7 Peer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor, School of Medicine: Psychiatry, Clinical, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005068
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: PTSD; Physical Injury
Keywords: PTSD; Physical Injury; Patient Concerns; Emergency Department Utilization
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-Integrated Multidisciplinary Collaborative Care (Experimental): The peer-integrated collaborative care intervention includes front-line trauma center staff (e.g., nursing and masters in social work), joined by injured peer interventionists and supervised by an MD (psychiatrist). The collaborative care team will provide case management, behavioral intervention elements, psychopharmacologic medication recommendations as well as 24/7 cell phone coverage for approximately 6 months post-injury. The intervention will be supported by a novel emergency department health information technology platform.
  Interventions: Behavioral: Peer-Integrated Multidisciplinary Collaborative Care
- Trauma surgery team notification (Active Comparator): Trauma surgery team notification of patient emotional distress, with recommendation for mental health inpatient consultation will be the comparator condition.
  Interventions: Behavioral: Trauma surgery team notification

INTERVENTIONS:
Behavioral: Peer-Integrated Multidisciplinary Collaborative Care — Case management, behavioral intervention elements, psychopharmacologic medication recommendations and 24/7 cell phone coverage for 6 months post-injury.
  Arms: Peer-Integrated Multidisciplinary Collaborative Care
Behavioral: Trauma surgery team notification — Trauma surgery team notification of patient emotional distress, with plan for mental health inpatient consultation will be the comparator condition.
  Arms: Trauma surgery team notification

SUMMARY:
This study evaluates two readily implementable approaches to the delivery of transitional care for injured patients treated emergently in US trauma care systems. The two approaches to be compared are a multidisciplinary team collaborative care intervention that integrates front-line trauma center staff with peer interventionists to trauma surgical team notification of patient emotional distress with recommended mental health consultation. The collaborative care intervention will be supported by a novel Emergency Department (ED) health information exchange technology platform.

DETAILED DESCRIPTION:
Collaborative care models are an established standard of care for treating combined mental health and chronic medical conditions in acute and primary care medical settings. However, very few interventions exist for the acute injury population transitioning between settings. While peer interventionist programs have been instituted for care delivery in many conditions, they have not yet been comprehensively integrated into acute post-injury interventions. Literature reviews support the need for comparative effectiveness trials of health care system interventions targeting high need injured patients with multiple complex mental health and medical comorbidities who are at risk for fragmented post-injury health service utilization. This study evaluates two readily implementable approaches to the delivery of transitional care for injured patients treated emergently in US trauma care systems. The two approaches to be compared are a multidisciplinary team collaborative care intervention that integrates front-line trauma center staff with peer interventionists to trauma surgical team notification of patient emotional distress with recommended mental health consultation. The collaborative care intervention will be supported by a novel Emergency Department (ED) health information exchange technology platform.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient/emergency admission for intentional and/or unintentional injury
* Score of ≥35 on the PTSD checklist
* Endorsement of ≥ 1 severe posttraumatic concern

Exclusion Criteria:

* Patients who required immediate psychiatric intervention
* Patients who are not Washington or Oregon State residents
* Patients who are currently incarcerated
* Patients not speaking Spanish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington Harborview Level I Trauma Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Palinkas LA, Engstrom A, Knutsen T, Walen ML, Whiteside L, Nehra D, Zatzick D. Implementation of a Face-To-Face Vs Virtual Peer-Integrated Collaborative Care Intervention for Mental Health Treatment of Physical Trauma Survivors: A Qualitative Study of Lessons from the COVID-19 Pandemic. Psychiatry. 2025 Nov 25:1-7. doi: 10.1080/00332747.2025.2592725. Online ahead of print. PMID 41289309
- [Derived] Iles-Shih M, Kelly G, McManamen M, Buggaveeti AE, Bulger E, Ryan P, Conde C, Huynh M, Ahmad M, Russo J, Wang J, Zatzick D. Can screening and referral for posttraumatic stress improve mental health and substance abuse service delivery at trauma centers? Results from a randomized trial. Injury. 2026 Jan;57(1):112845. doi: 10.1016/j.injury.2025.112845. Epub 2025 Oct 25. PMID 41173731
- [Derived] Zatzick DF, Bulger EM, Thomas P, Engstrom A, Iles-Shih M, Russo J, Wang J, Shoyer J, Conde C, Abu K, Birk N, Palinkas L, Heagerty P, Whiteside LK, Ryan P, Knutzen T, Maier R. Randomized clinical trial of peer integrated collaborative care intervention after physical injury. Trauma Surg Acute Care Open. 2025 Jan 19;10(1):e001657. doi: 10.1136/tsaco-2024-001657. eCollection 2025. PMID 39845998
- [Derived] Scheuer H, Engstrom A, Thomas P, Moodliar R, Moloney K, Walen ML, Johnson P, Seo S, Vaziri N, Martinez A, Maier R, Russo J, Sieber S, Anziano P, Anderson K, Bulger E, Whiteside L, Heagerty P, Palinkas L, Zatzick D. A comparative effectiveness trial of an information technology enhanced peer-integrated collaborative care intervention versus enhanced usual care for US trauma care systems: Clinical study protocol. Contemp Clin Trials. 2020 Apr;91:105970. doi: 10.1016/j.cct.2020.105970. Epub 2020 Feb 29. PMID 32119926

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peer-Integrated Multidisciplinary Collaborative Care | Trauma Surgery Team Notification
Started | 225 | 225
Completed | 225 | 225
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer-Integrated Multidisciplinary Collaborative Care | Trauma Surgery Team Notification | Total
Number analyzed (Participants) | 225 | 225 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (15.1) | 38.5 (15.5) | 38.9 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 109 | 220
  Male | 114 | 116 | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 53 | 109
  Not Hispanic or Latino | 168 | 172 | 340
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 6 | 20
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 5 | 3 | 8
  Black or African American | 38 | 32 | 70
  White | 112 | 125 | 237
  More than one race | 29 | 26 | 55
  Unknown or Not Reported | 22 | 29 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With 1 or More Emergency Department Visits Per Quarter
Description: Number of emergency visits will be assessed using the Emergency Department Information Exchange (EDIE). More emergency visits are indicative of a worse outcome.
Time Frame: Baseline injury admission to 12-months post-injury follow-up
Population: For the number of emergency department visits outcome, electronic health record data accrued on the entire intent-to-treat sample (N = 450) over the course of the 12-months after injury hospitalization. Mixed-model regression analyses will be incorporated into the data analytic approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer-Integrated Multidisciplinary Collaborative Care | Trauma Surgery Team Notification
Number analyzed (Participants) | 225 | 225
Participants
  Baseline | 225 | 225
  First Quarter | 90 | 79
  Second Quarter | 52 | 38
  Third Quarter | 49 | 50
  Fourth Quarter | 47 | 40

2. Primary Outcome: Change in Posttraumatic Concern Severity
Description: The severity of patient described post-injury concerns as rated by patients on a 1 through 5 scale; 1 being not at all concerning and 5 being extremely concerning. Higher scores are indicative of a worse outcome. The concern outcome can either be represented as a mean severity score or as a percentage of patients with one or more severe concerns.
Time Frame: Baseline injury admission and 1-, 3-, 6-, 9- and 12-months post-injury follow-up
Population: For the severity of patient described post-injury concerns outcome, self-report data was collected from individual patients at each time point. Patient self-report interview follow-up completion varied at each time point across the intervention and control conditions. This accounts for samples less than 225 at the 1-, 3-, 6- , 9- and 12-month time points. Mixed-model regression analyses will be incorporated into the data analytic approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer-Integrated Multidisciplinary Collaborative Care | Trauma Surgery Team Notification
Number analyzed (Participants) | 225 | 225
Participants
  Baseline | 225 | 225
  1 month: number analyzed (Participants) | 206 | 194
  1 month | 152 | 140
  3 month: number analyzed (Participants) | 190 | 188
  3 month | 130 | 133
  6 month: number analyzed (Participants) | 180 | 161
  6 month | 129 | 97
  9 month: number analyzed (Participants) | 171 | 154
  9 month | 101 | 100
  12 month: number analyzed (Participants) | 180 | 167
  12 month | 111 | 95

3. Primary Outcome: Change in Posttraumatic Stress Disorder (PTSD) Symptoms
Description: The investigators will use the PTSD Checklist - Civilian (PCL-C). The scoring of the scale ranges from a minimum of 17 to a maximum of 85, with higher scores indicating a worse outcome. The measure can also provide a rating of symptoms consistent with a diagnosis of PTSD.
Time Frame: Baseline injury admission and 1-, 3-, 6-, 9- and 12-months post-injury follow-up
Population: For the posttraumatic stress symptom outcome, self-report data was collected from individual patients at each time point. Patient self-report interview follow-up completion varied at each time point across the intervention and control conditions. This accounts for samples less than 225 at the 1-, 3-, 6- , 9- and 12-month time points. Mixed-model regression analyses will be incorporated into the data analytic approach.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer-Integrated Multidisciplinary Collaborative Care | Trauma Surgery Team Notification
Number analyzed (Participants) | 225 | 225
units on a scale
  Baseline | 49.3 (11.3) | 49.5 (11.4)
  1 month: number analyzed (Participants) | 206 | 193
  1 month | 44.0 (15.8) | 44.1 (16.4)
  3 month: number analyzed (Participants) | 190 | 187
  3 month | 40.2 (15.4) | 42.6 (16.4)
  6 month: number analyzed (Participants) | 182 | 160
  6 month | 40.2 (16.0) | 40.8 (15.8)
  9 month: number analyzed (Participants) | 170 | 154
  9 month | 39.9 (15.0) | 40.7 (16.8)
  12 month: number analyzed (Participants) | 180 | 168
  12 month | 38.6 (15.7) | 39.8 (17.1)

4. Primary Outcome: Change in Functional Status
Description: The investigators will use the Medical Outcomes Study Short Form healthy survey (MOS Short Form-12/36) physical components summary to assess physical function. The minimum and maximum scores are 0-100 with higher scores representing a better outcome.
Time Frame: Baseline injury admission and 1-, 3-, 6-, 9- and 12-months post-injury follow-up
Population: For the physical functional status outcome, self-report data was collected from individual patients at each time point. Patient self-report interview follow-up completion varied at each time point across the intervention and control conditions. This accounts for samples less than 225 at the 1-, 3-, 6- , 9- and 12-month time points. Mixed-model regression analyses will be incorporated into the data analytic approach.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer-Integrated Multidisciplinary Collaborative Care | Trauma Surgery Team Notification
Number analyzed (Participants) | 225 | 225
units on a scale
  Baseline | 49.4 (11.1) | 50.2 (10.3)
  1 month: number analyzed (Participants) | 200 | 191
  1 month | 31.0 (6.8) | 30.0 (7.5)
  3 month: number analyzed (Participants) | 186 | 185
  3 month | 35.4 (10.2) | 33.7 (10.4)
  6 month: number analyzed (Participants) | 179 | 152
  6 month | 37.4 (12.1) | 36.9 (9.9)
  9 month: number analyzed (Participants) | 165 | 152
  9 month | 38.4 (11.3) | 37.9 (11.1)
  12 month: number analyzed (Participants) | 172 | 159
  12 month | 39.8 (12.3) | 39.2 (11.1)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the year after injury hospitalization.
Arm/Group | Peer-Integrated Multidisciplinary Collaborative Care | Trauma Surgery Team Notification
All-Cause Mortality (participants affected / at risk) | 6/225 | 4/225
Serious Adverse Events (participants affected / at risk) | 13/225 | 7/225
Other Adverse Events (participants affected / at risk) | 119/225 | 117/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peer-Integrated Multidisciplinary Collaborative Care (N=225) | Trauma Surgery Team Notification (N=225)
Presentation to emergency department with suicidal ideation or intent (Psychiatric disorders) | 7 | 3
Death (Injury, poisoning and procedural complications) | 6 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peer-Integrated Multidisciplinary Collaborative Care (N=225) | Trauma Surgery Team Notification (N=225)
Suicidal Ideation (Psychiatric disorders) | 119 | 117 — Suicidal ideation reported on the Patient Health Questionnaire Nine Item Survey, Item 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT03569878/Prot_SAP_000.pdf